CLINICAL TRIAL: NCT03953560
Title: Symptom-related Screening Program Following Pulmonary Embolism for Early Detection of Chronic ThromboEmbolic Pulmonary Hypertension (CTEPH)
Brief Title: Symptom-related Screening for Early Detection of CTEPH.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Luis Jara-Palomares, MD (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry); Sociedad Española de Neumología y Cirugía Torácica (Other)
Responsible Party: Sponsor-Investigator, Luis Jara-Palomares, MD, Principal Investigator, Hospitales Universitarios Virgen del Rocío
Organization: Hospitales Universitarios Virgen del Rocío (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 0034667956480
Record Dates: First submitted 2019-05-14; First posted 2019-05-16 (Actual); Last update posted 2022-03-17 (Actual); Status verified 2022-03

CONDITIONS: CTEPH; Pulmonary Embolism; Symptoms and Signs; Dyspnea
Keywords: CTEPH; Pulmonary Embolism; Symptoms and Signs; Dyspnea
MeSH Terms: conditions — Pulmonary Embolism; Signs and Symptoms; Dyspnea

STUDY DESIGN:
Intervention Model Description: Design Cohorts study in consecutive patients with objectively confirmed PE.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Screening (Experimental): Intervention Investigator from each center will recover consecutives PE patients and collect baseline, demographic and comorbidities.
  In all patients enrolled in the study a short questionnaire regarding dyspnea symptoms will be performed. All patients that refer dyspnea grade ≥ II according NYHA-WHO (6) modified scale will be cited as outpatient to be evaluated Imaging studies and right heart catheterization is the procedure agreeing with the standard care according to current ESC/ERS Guidelines.
  In all patients, the following tests will be performed:
  1. Pulsioximetry.
  2. Electrocardiogram.
  3. Blood sample with determination of NT-ProBNP.
  4. Echocardiography. Only an echocardiography indicative of PH warrants further evaluation
  5. V/Q scintigraphy. Possible CTEPH can be assumed when mismatched perfusion defects are detected by VQ scan.
  6. Right heart catheterization & Pulmonary CT Scan are required for confirming the diagnosis
  Interventions: Diagnostic Test: dyspnea grade ≥ II according NYHA-WHO

INTERVENTIONS:
Diagnostic Test: dyspnea grade ≥ II according NYHA-WHO — Intervention Investigator from each center will recover consecutives PE patients and collect baseline, demographic and comorbidities.
  In all patients enrolled in the study a short questionnaire regarding dyspnea symptoms will be performed. All patients that refer dyspnea grade ≥ II according NYHA-WHO (6) modified scale will be cited as outpatient to be evaluated
  Imaging studies and right heart catheterization is the procedure agreeing with the standard care according to current ESC/ERS Guidelines.
  In all patients, the following tests will be performed:
  1. Pulsioximetry.
  2. Electrocardiogram.
  3. Blood sample with determination of NT-ProBNP.
  4. Echocardiography. Only an echocardiography indicative of PH warrants further evaluation
  5. V/Q scintigraphy. Possible CTEPH can be assumed when mismatched perfusion defects are detected by VQ scan.
  6. Right heart catheterization & Pulmonary CT Scan are required for confirming the diagnosis

SUMMARY:
Routine screening for Chronic thromboembolic pulmonary hypertension (CTEPH) i after PE is not supported by current evidence and guidelines.

This study aims to evaluate if a screening program for patients with acute PE based on telephone monitoring of symptoms and further examination if only symptomatic patients could help an early detection of CTEPH.

DETAILED DESCRIPTION:
Chronic thromboembolic pulmonary hypertension (CTEPH) is a long-term complication following an acute or silent pulmonary embolism (PE). A history of acute PE was reported in 75% of CTEPH patients. Nevertheless, incidence of CTEPH after a confirmed acute PE vary widely depending of the studies, with estimated incidence from 0.5 to 4%. Performing a follow-up examination of patients diagnosed with acute PE regardless of persisting symptoms and using all available technical procedures is not cost-effective. As a consequence, routine screening for CTEPH after PE is not supported by current evidence and guidelines.

CTEPH is a very disabling and mortal disease, although it is a potential curable disease. However, delayed diagnosis and misdiagnosis is common. Patients are frequently diagnosed with CTEPH at advanced stages of the disease leading to worse clinical outcomes. Early diagnosis of CTEPH is essential, as delay in diagnosis may be associated with a worse prognosis, higher perioperative mortality and inoperable diseases stages. Overall, evidence from various sources suggests that early detection and treatment of CTEPH is advantageous in achieving favorable clinical outcomes. Therefore, there is an important unmet need for early diagnosing this disease.

Focusing diagnostic procedures only on symptomatic patients may be a practical approach for detecting relevant CTEPH.

This study aims to evaluate if a screening program for patients with acute PE based on telephone monitoring of symptoms and further examination if only symptomatic patients could help an early detection of CTEPH.

Objectives

* Primary outcome: To estimate the impact of an easy and simple strategy to identify CTEPH.
* Secondary outcomes:

  * To identify patients with CTED after PE
  * To obtain external validation from scores to identify patients at risk to develop CTEPH
  * To develop new score to identify high risk population to develop CTEPH

Hypothesis Conceptual hypothesis: The use of a strategy to detect CTEPH will increase number of patients diagnosed of pulmonary hypertension.

Operational hypothesis: The use of a strategy to detect CTEPH will increase in a 200% the number of patients diagnosed with CTEPH.

Design Cohorts study in consecutive patients with objectively confirmed PE.

Specialists implied Internal medicine, Pulmonologist, Hematologist from 20 hospitals.

Inclusion criteria: 1) Age > 18 year 2) Objectively confirmed diagnosis of acute PE by multidetector CT, V/Q lung scan, or selective pulmonary angiography, according to established diagnostic criteria, with or without symptomatic DVT, 3) Ability of subject to understand the character and consequences of the study, 4) informed consent of the subject. Exclusion criteria: refused informed consent, inability to cooperation.

Intervention Investigator from each center will recover consecutive PE patients and collect baseline, demographic and co-morbidities.

In all patients enrolled in the study a short questionnaire regarding dyspnea symptoms will be performed. All patients that refer dyspnea grade ≥ II according NYHA-WHO modified scale will be cited as outpatient to be evaluated

A written informed consent will be required all patients evaluated in consultant.

Imaging studies and right heart catheterization is the procedure agreeing with the standard care according to current ESC/ERS Guidelines.

In all patients, the following tests will be performed:

1. Pulsioximetry.
2. Electrocardiogram.
3. Blood sample with determination of NT-ProBNP.
4. Echocardiography. Only an echocardiography indicative of PH warrants further evaluation
5. V/Q scintigraphy. Possible CTEPH can be assumed when mismatched perfusion defects are detected by VQ scan.
6. Right heart catheterization & Pulmonary CT Scan are required for confirming the diagnosis

The relationship of Doppler echocardiography-estimated PASP with right heart catheterization (RHC)-measured PASP was examined using Spearman's correlation coefficients. The Bland-Altman method was then used to assess the agreement between Doppler echocardiography-estimated and RHC measured PASP. Doppler echocardiography-estimated PASP within +/- 10mmHg of the value measured on RHC was considered accurate, consistent with the cutoffs used in other publications.

Secondary outcome include number of patients with chronic thromboembolic disease (CTED), described as chronic thromboembolic pulmonary vascular obstruction with normal resting pulmonary artery pressures.

Treatment: No treatment required

Statistical Plans Sample size calculation We estimate CTEPH prevalence in reference group of 1%, and a prevalence of CTEPH in interventional group of 2.8%. With unilateral test, con confidence level of 95%, statistic power of 80% and losses expected of 25%, we calculated a final sample size of 947.

The investigators calculate that 16-20 centers in Spain are needed to recruit patients

Investigators will compare baseline characteristics of patients with and without CTEPH using chi-square tests for categorical variables and non-parametric rank tests for continuous variables. Cumulative incidence of CTEPH will be estimated using the Kaplan-Meier technique.

To do external validation of previous score to predict CTEPH discriminative power by calculating the area under the receiver-operating characteristic (ROC) curve will be done, performing a non-parametric test of the equality of the areas under the ROC curves. Goodness-of-fit of the score points for each score in a logistic regression model using Pearson's chi-square test.

Student's t test and X2 test (or Fisher's exact test where appropriate) will be used to compare continuous or categorical variables, and multivariable analysis through a logistic regression model using the Wald method (step back) to identify independent predictors for the occurrence of CTEPH. Covariates entering in the model will be selected by a significance level of p <0.20 on univariable analysis, or by a well-known association reported in the literature. Then, the investigators will build a prognostic score assigning points to each independent variable according to regression coefficients β, rounding to the nearest integer. The investigators will assign a risk score to each patient by adding up points for each independent variable. Performance will be quantified in terms of calibration using the Hosmer-Lemeshow test. Model discrimination will be assessed using the C-statistic. Internal validity of the score will be confirmed using bootstrap analysis. For the statistical analysis the investigators will use the IBM SPSS Statistics program (version 19; SPSS Inc., Chicago, IL), and a two-sided p<0.05 was considered to be statistically significant.

ELIGIBILITY:
Inclusion Criteria:

1. Age > 18 year
2. Objectively confirmed diagnosis of acute PE by multidetector CT, V/Q lung scan, or selective pulmonary angiography, according to established diagnostic criteria, with or without symptomatic DVT,
3. Ability of subject to understand the character and consequences of the study,
4. informed consent of the subject.

Exclusion Criteria:

* refused informed consent, inability to cooperation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 646 (Actual)
Dates: Start 2019-01-16 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2022-02-15 (Actual)

PRIMARY OUTCOMES:
Number of new diagnosis of CTEPH | Up 3 years after PE
  New diagnosis of CTEPH

SECONDARY OUTCOMES:
External validation from score to identify patients at risk to develop CTEPH | Up 3 years after PE
  external validation from score (Klok FA et al. Derivation of a clinical prediction score for chronic thromboembolic pulmonary hypertension after acute pulmonary embolism. J Thromb Haemost. 2016)
Derivation of a score to identify high risk population to develop CTEPH | Up 3 years after PE
  With variables assocciated to CTEPH investigators will obtain derivation and validation of a score to identify high risk population to develop CTEPH
Number of patients with Chronic Thromboembolic Disease (CTED) after PE | Up 3 years after PE
  Describe the number and clinical characteristics of patients with CTED after PE

CONTACTS AND LOCATIONS:
Overall Officials: Luis Jara-Palomares, MD, Study Director — Medical Surgical Unit of Respiratory Diseases, Virgen del Rocio Hospital, CIBERES
Locations (16):
- Spain (16):
  - Hospital Universitario Puerto Real, Puerto Real, Cadiz
  - Consorcio Hospitalario Provincial de Castellón, Castellon, Castellon
  - Hospital de Galdakao, Galdakao, Vizcaya
  - Hospital General Universitario de Albacete, Albacete
  - Hospital Universitario de Bellvitge, Barcelona
  - Parc Sanitari Sant Joan de Deu, Barcelona
  - Hospital Universitario Reina Sofía, Córdoba
  - Hospital Virgen de la Luz, Cuenca
  - Hospital General Universitario de Elche, Elche
  - Hospital Universitari de Girona Dr. Josep Trueta, Girona
  - Hospital Universitari Arnau de Vilanova, Lleida
  - Hospital Clínico San Carlos, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Virgen del Rocio, Seville
  - Hospital Universitario Joan XXIII de Tarragona, Tarragona
  - Hospital Clínico Universitario Lozano Blesa, Zaragoza

IPD SHARING:
Plan to Share IPD: No
Data will be included in RIETE registry. We will done all analyses prestablished and data collected could be used by RIETE investigators

REFERENCES:
- [Derived] Marin-Romero S, Ballaz-Quincoces A, Gomez-Cuervo C, Marchena-Yglesias PJ, Lopez-Miguel P, Francisco-Albesa I, Pedrajas-Navas JM, Lumbierres M, Aibar-Arregui MA, Bosco Lopez-Saez J, Perez-Pinar M, Baeza-Martinez C, Riera-Mestre A, Peris-Sifre M, Porras-Ledantes JA, Criado-Garcia J, Elias-Hernandez T, Otero R, Barca-Hernando M, Muriel A, Klok FA, Jara-Palomares L; SYSPPE investigators. Symptom-related screening programme for early detection of chronic thromboembolic pulmonary hypertension after acute pulmonary embolism: the SYSPPE study. Thorax. 2024 Jan 18;79(2):144-152. doi: 10.1136/thorax-2023-220580. PMID 38050187